CLINICAL TRIAL: NCT06661083
Title: Counteracting HPV Infection with Natural Molecules
Brief Title: The Effect of Natural Molecules on HPV Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AGUNCO Obstetrics and Gynecology Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Epistop_2024
Record Dates: First submitted 2024-10-23; First posted 2024-10-28 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: HPV (Human Papillomavirus)-associated
MeSH Terms: conditions — Papillomavirus Infections | interventions — epigallocatechin gallate; Vitamin B 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with HPV infection (Experimental)
  Interventions: Dietary Supplement: EGCG, FA, HA, B12

INTERVENTIONS:
Dietary Supplement: EGCG, FA, HA, B12 — EGCG + FA + HA + B12 (1 cps /die)

SUMMARY:
The purpose of the study is to evaluate the effect of the administration of natural molecules in the treatment of HPV infection.

ELIGIBILITY:
Inclusion Criteria:

* HPV DNA test positivity
* over 18 years

Exclusion Criteria:

* pregnancy
* breastfeeding
* assumption of other products containing EGCG or green tea
* primary immunodepression or pharmacological induced one

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-03-07 (Actual)

PRIMARY OUTCOMES:
HPV DNA test negativity | 6 months of treatment
  Percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Agunco, Rome, Italy